CLINICAL TRIAL: NCT02571517
Title: Impact of the Administration of Systemic Glucocorticoids on Inflammatory Response and Clinical Evolution of Patients Diagnosed With Moderate- Severe Bronchiolitis
Brief Title: Glucocorticoid Therapy Impact on the Inflammatory Response and Clinical Evolution in Patients With Severe Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSJD-GLUCOBR-2010; 2011-000337-36 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Bronchiolitis, Viral
Keywords: Respiratory viral infection.; Respiratory syncytial virus bronchiolitis; METHYLPREDNISOLONE SODIUM SUCCINATE
MeSH Terms: conditions — Bronchiolitis, Viral | interventions — Glucocorticoids; Methylprednisolone; Methylprednisolone Hemisuccinate; Glucose; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucocorticoids (Experimental): methylprednisolone intravenous administration of 2mg/kg/day (divided in two doses) and/or oral prednisolone 2,5 mg/kg/day (in two divided doses) during 7 days.
  Patients younger than 2 year, who required hospitalization, affected by moderate or severe bronchiolitis
  Interventions: Drug: Glucocorticoids
- Placebo (Placebo Comparator): will receive iv/oral glucose 5% solution as placebo of 2mg/kg/day and/or 2,5 mg/kg/day (divided in two doses) during 7 days.
  Patients younger than 2 year, who required hospitalization, affected by moderate or severe bronchiolitis.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glucocorticoids — Patients assigned to experimental group (group 1) will receive iv methylprednisolone 2 mg/kg/day (divided in two doses) doses and/or oral prednisolone 2,5 mg/kg/day (divided in two doses) during 7 days.
  Other Names: SOLU-MODERIN 125 mg; METHYLPREDNISOLONE SODIUM SUCCINATE; ESTILSONA Gotas
  Arms: Glucocorticoids
Other: Placebo — Patients assigned to control group (group 2) will receive iv/oral glucose 5% solution as placebo, 2 mg/kg/day (divided in two doses) during 7 days.
  Other Names: glucose 5% solution; Plast-Apyr Glucosado 5%
  Arms: Placebo

SUMMARY:
The purpose of this study is to to demonstrate that a 7-day course of systemic glucocorticoids decreases the inflammatory activity of moderate or severe bronchiolitis in paediatric patients compared to the standard treatment. To evaluate the morbidity (regarding to the clinical course: Intensive Pediatric Unit Care unit (PICU) admission, mechanical ventilation, ionotropic support, nosocomial infection, rescue therapy for respiratory failure; duration of PICU stay and hospitalization; and exitus) between the treatment and the control groups.

DETAILED DESCRIPTION:
A Prospective, randomised, double blind and placebo controlled study. Patients assigned to experimental group (group 1) will receive iv methylprednisolone 2 mg/kg/day (in two divided doses) and/or oral prednisolone 2,5 mg/kg/day (in two divided doses) every 12 hours, during 7 days.

Patients assigned to control group (group 2) will receive iv/oral glucose 5% solution as placebo, at the same dose and time as the experimental group. A total of 50 (initially 39, but it was extended to 50 by Protocol Amendment) patients per group are recruited.

Bronchiolitis is the most common infection of the lower respiratory tract. It is defined as, the first episode of bronchospasm, dyspnea, expiratory difficulty, feed refusal, tachypnea greater than 50 rpm and radiological evidence of hyperinflation, in less than 24 months.

It is a very prevalent disease, Respiratory syncytial virus (RSV) infects 70% of children under one year and 100% of children under 2 years and generates a major health impact on epidemic period (especially from December to February) . It is the most frequent cause of hospitalization in children under one year during the winter and up to 10% of those admitted will need intensive care, of which up to 60% required intubation and mechanical ventilation. The estimated disease in healthy children, mortality ranges from 0.005% to 0.02%, while in hospitalized children becomes between 1% and 3%.

In recent years, there have been numerous studies, mainly in RSV bronchiolitis, to analyze the immunological basis of the disease, as discussed complex, in order to perform a prophylaxis and treatment of more optimal infection.

Inflammatory response in bronchiolitis results in activation of cytokines and chemokines that generates a viral clearance. However, if the inflammatory response is disproportionate, the pathogenesis of the disease can lead to a worse clinical evolution.

Corticosteroids are drugs having inhibitory effects on specific immune response, mediated both T cells and the B cell, and are potent inhibitors of phagocyte function. These drugs are effective in the management of multiple forms of secondary inflammatory diseases or immune disorders and may also be useful in the management of bronchiolitis.

The treatment of bronchiolitis is mainly based on supportive therapy: oxygen therapy, proper hydration and aspiration of nasal secretions. Many treatments have been tried that have tried to lessen the severity of the infection, such as the use of bronchodilators and / or corticosteroids, although with controversial results.

In the literature review conducted in PubMed, the investigators found about 110 related bronchiolitis, as MeSH Terms, publications using the words "bronchiolitis" [All Fields] AND ("child" [MeSH Terms].

Only three of these articles shows results of clinical trials, although none in relation to the usefulness of steroids in bronchiolitis.

There is just a case report describing the use of intravenous corticosteroids in infants with severe bronchiolitis, in combination with therapies such as extracorporeal oxygenation.

One of the important aspects that the investigators took in consideration is that rhinovirus bronchiolitis is one of the most involved cause in the development of asthma, and just one of the etiologies of bronchiolitis who could benefit from treatment with corticosteroids.

Prednisolone and methylprednisolone are also well known and used drugs, whose side effects are often dose and duration dependent.

The identification and recruitment of patients will take place during the admission in the Intensive Pediatric Unit Care unit at the Hospital Sant Joan de Deu.

Treatment of patients starts on days 0 and 3 of hospitalization. The patient treatment duration is 7 days, after that starts the follow-up phase, which duration is one month from the date of the baseline visit and until the hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

The study will recruit paediatric patients younger than one year old who require hospitalization for moderate-severe bronchiolitis according to the BRONCHIOLITIS SCORE of Sant Joan de Deu Hospital (HSJD)

Exclusion Criteria:

* Patients of either gender under one year old with mild bronchiolitis.
* Patients with bronchiolitis in which the principal symptom is apnoea.
* Patients who have received corticotherapy before admission to hospital.
* No consent from parents or tutors.
* Patients with previous acquired or innate immunodepression.
* Patients enrolled in other clinical trials.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in inflammatory response | enrollment to one week treatment
  inflammatory response evaluation of the first week of glucocorticoids treatment as assessed by multiple measurements aggregated to arrive at one reported value, which are: the bronchiolitis clinical severity Scale, pediatric mortality Risk scale (PRISM III), the Chest x-ray test, the nasopharyngeal aspiration and analytical exploration (at day 5-7)
Morbidity episodes | 14 months
  Morbidity assessment by multiple measurements aggregated to arrive at one reported value which are as follow: necessity of mechanical ventilation, inotropic, presence of nosocomial infection, rescue therapies if respiratory failure occur; days of admission to the Pediatric Intensive Care Unit and hospitalization, in both treatment and control groups

SECONDARY OUTCOMES:
Number of Side effects estimate | 14 months
  Number of Side effects estimate by comparing the experimental group to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Iolanda Jordán, MD, Principal Investigator — UCIP H Sant Joan de Déu

REFERENCES:
- [Background] Bonzel L, Tenenbaum T, Schroten H, Schildgen O, Schweitzer-Krantz S, Adams O. Frequent detection of viral coinfection in children hospitalized with acute respiratory tract infection using a real-time polymerase chain reaction. Pediatr Infect Dis J. 2008 Jul;27(7):589-94. doi: 10.1097/INF.0b013e3181694fb9. PMID 18520973
- [Background] Ogra PL. Respiratory syncytial virus: the virus, the disease and the immune response. Paediatr Respir Rev. 2004;5 Suppl A:S119-26. doi: 10.1016/s1526-0542(04)90023-1. PMID 14980256
- [Background] Harris JA, Huskins WC, Langley JM, Siegel JD; Pediatric Special Interest Group of the Society for Healthcare Epidemiology of America. Health care epidemiology perspective on the October 2006 recommendations of the Subcommittee on Diagnosis and Management of Bronchiolitis. Pediatrics. 2007 Oct;120(4):890-2. doi: 10.1542/peds.2007-1305. No abstract available. PMID 17908774
- [Background] Bueno SM, Gonzalez PA, Pacheco R, Leiva ED, Cautivo KM, Tobar HE, Mora JE, Prado CE, Zuniga JP, Jimenez J, Riedel CA, Kalergis AM. Host immunity during RSV pathogenesis. Int Immunopharmacol. 2008 Oct;8(10):1320-9. doi: 10.1016/j.intimp.2008.03.012. Epub 2008 Apr 14. PMID 18687294
- [Background] Chatham WW, Kimberly RP. Treatment of lupus with corticosteroids. Lupus. 2001;10(3):140-7. doi: 10.1191/096120301675075008. PMID 11315342
- [Background] Jat KR, Chawla D. Surfactant therapy for bronchiolitis in critically ill infants. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD009194. doi: 10.1002/14651858.CD009194.pub2. PMID 22972138